CLINICAL TRIAL: NCT01012297
Title: A Randomized Phase III Evaluation of Docetaxel (NSC #628503) and Gemcitabine (NSC #613327) Plus G-CSF With Bevacizumab (NSC #704865) Versus Docetaxel (NSC #628503) and Gemcitabine (NSC #613327) Plus G-CSF With Placebo in the Treatment of Recurrent or Advanced Leiomyosarcoma of the Uterus
Brief Title: Gemcitabine Hydrochloride and Docetaxel With or Without Bevacizumab in Treating Patients With Advanced or Recurrent Uterine Leiomyosarcoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was targeted to accrue 130 patients, but closed early for futility.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2010-01738; NCI-2010-01738 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000659024; GOG-0250; GOG-0250 (Other: NRG Oncology); GOG-0250 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Recurrent Uterine Corpus Sarcoma; Stage IIIA Uterine Sarcoma; Stage IIIB Uterine Sarcoma; Stage IIIC Uterine Sarcoma; Stage IVA Uterine Sarcoma; Stage IVB Uterine Sarcoma; Uterine Corpus Leiomyosarcoma
MeSH Terms: interventions — Bevacizumab; Immunoglobulin G; Disulfides; Docetaxel; Filgrastim; Granulocyte Colony-Stimulating Factor; Gemcitabine; pegfilgrastim

ARMS (2):
- Arm I Gem+Doce+Placebo (Experimental): Patients receive a placebo IV over 30-90 minutes on day 1, gemcitabine hydrochloride IV over 90 minutes on days 1 and 8, and docetaxel IV over 60 minutes on day 8. Patients also receive filgrastim subcutaneously (SC) on days 9-15 or pegfilgrastim SC on day 9 or 10.
  Interventions: Drug: Docetaxel; Biological: Filgrastim; Drug: Gemcitabine Hydrochloride; Biological: Pegfilgrastim; Other: Placebo
- Arm II Gem+Doce+Bev (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1, gemcitabine hydrochloride IV over 90 minutes on days 1 and 8, and docetaxel IV over 60 minutes on day 8. Patients also receive filgrastim SC on days 9-15 or pegfilgrastim SC on day 9 or 10.
  Interventions: Biological: Bevacizumab; Drug: Docetaxel; Biological: Filgrastim; Drug: Gemcitabine Hydrochloride; Biological: Pegfilgrastim

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm II Gem+Doce+Bev
Drug: Docetaxel — Given IV
  Other Names: RP56976; Taxotere; Taxotere Injection Concentrate
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Neulasta; SD-01; SD-01 sustained duration G-CSF
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm I Gem+Doce+Placebo

SUMMARY:
This randomized phase III trial is studying gemcitabine hydrochloride, docetaxel, and bevacizumab to see how well they work compared with gemcitabine hydrochloride, docetaxel, and a placebo in treating patients with advanced or recurrent uterine leiomyosarcoma. Drugs used in chemotherapy, such as gemcitabine hydrochloride and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether gemcitabine hydrochloride and docetaxel are more effective when given with or without bevacizumab in treating uterine leiomyosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of bevacizumab to fixed-dose rate gemcitabine-docetaxel reduces the progression-free survival (PFS) event rate when compared to gemcitabine-docetaxel plus placebo in patients with advanced or recurrent uterine leiomyosarcoma (LMS).

SECONDARY OBJECTIVES:

I. To determine the objective response rate, as measured by RECIST, of patients treated with fixed-dose rate gemcitabine-docetaxel with bevacizumab, compared with the objective response rate of patients treated with fixed-dose rate gemcitabine-docetaxel with placebo.

II. To determine if the addition of bevacizumab to the combination of gemcitabine and docetaxel increases overall survival in patients with advanced or recurrent uterine LMS.

III. To determine the toxicity profile of fixed-dose rate gemcitabine-docetaxel with and without bevacizumab in this patient population.

IV. To bank formalin-fixed and paraffin-embedded (FFPE) tumor tissue for research.

OUTLINE: This is a multicenter study. Patients are stratified according to prior whole-pelvic radiotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive a placebo IV over 30-90 minutes on day 1, gemcitabine hydrochloride IV over 90 minutes on days 1 and 8, and docetaxel IV over 60 minutes on day 8. Patients also receive filgrastim subcutaneously (SC) on days 9-15 or pegfilgrastim SC on day 9 or 10.

ARM II: Patients receive bevacizumab IV over 30-90 minutes on day 1, gemcitabine hydrochloride IV over 90 minutes on days 1 and 8, and docetaxel IV over 60 minutes on day 8. Patients also receive filgrastim SC on days 9-15 or pegfilgrastim SC on day 9 or 10.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced or recurrent uterine leiomyosarcoma with documented disease progression; histologic confirmation of the original primary tumor is required
* All patients must have measurable disease as defined by RECIST 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patient must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must have a GOG Performance Status of 0, 1, or 2
* Patients must have recovered from effects of recent surgery, radiotherapy or other therapy
* Patients should be free of active infection requiring antibiotics (with the exception of an uncomplicated UTI)
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to first day of study treatment; continuation of hormone replacement therapy is permitted
* Platelet count greater than or equal to 100,000/mm^3
* ANC count greater than or equal to 1,500/mm^3
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), per NCI CTCAE Version 4.0 Grade 1
* Bilirubin within normal range (CTCAE Version 4 Grade 0)
* SGOT and alkaline phosphatase less than or equal to 2.5 x ULN, per the CTCAE Version 4.0 Grade 1)
* SGOT less than or equal to 2.5 x ULN, per the CTCAE Version 4.0 Grade 1
* Alkaline phosphatase less than or equal to 2.5 x ULN, per the CTCAE Version 4.0 Grade 1
* Neuropathy (sensory and motor) less than or equal to Grade 1 per the CTCAE Version 4.0.
* No history of transient ischemic attack (TIA) or stroke or CNS hemorrhage within the past 6 months
* Urine protein creatinine (UPC) ratio must be < 1.0 gm; if UPC ratio >= 1, collection of 24-hour urine measurement of urine protein is recommended
* PT such that international normalized ratio (INR) is =< 1.5 and a PTT =< 1.5 times the institutional upper limit of normal (or an in-therapeutic-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin)
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception

Exclusion Criteria:

* Patients who have received prior cytotoxic chemotherapy for management of uterine sarcoma; patients who have received prior VEGF-pathway targeted agent such as bevacizumab, PTK787, VEGF-trap, or who have received prior treatment with a multi-kinase inhibitor such as sorafenib or sunitinib are not eligible
* Patients who have had prior therapy with docetaxel or gemcitabine or bevacizumab
* Patients with a history of other invasive malignancies, with the exceptions of non-melanoma skin cancer, carcinoma in situ of the cervix, and ductal carcinoma in situ of the breast, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels; (necessary use of warfarin or low molecular weight heparin is permitted, provided the INR is maintained in the therapeutic range of approximately 2-3)
* Patients with major surgery or significant traumatic injury within 28 days prior to study entry
* Patients with a history of abdominal fistula or perforation within the past 12 months
* Patients with a current, serious, non-healing wound, ulcer, or bone fracture
* Patients with history or evidence upon physical examination of CNS disease, including history of primary brain tumor, or any history of brain metastases, or seizures not controlled with standard medical therapy
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Cardiovascular function; specifically, patient may not have:

  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 100 mm Hg in a patient with no history of hypertension; patients with a history of hypertension before enrollment on study are permitted, but such patients must have BP less than or equal to 140/90 mmHg; use of blood pressure medications to achieve and maintain blood pressure control is permitted
  * Myocardial infarction or unstable angina within 6 months of the first date of bevacizumab/placebo therapy
  * New York Heart Association (NYHA) Grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication; women who have received prior treatment with an anthracycline (including doxorubicin and/or liposomal doxorubicin) and have an ejection fraction < 50% will be excluded from the study
  * Grade 1, Category 2 or greater, peripheral vascular disease; patient cannot have anything worse than mild, symptomatic claudication with exercise
  * History of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of bevacizumab/placebo therapy
  * History of pulmonary embolism or deep vein thrombosis in the past 6 months
* Patients with, or with anticipation of, invasive procedures as defined below:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of bevacizumab/placebo therapy
  * Major surgical procedure anticipated during the course of the study.
  * Minor surgical procedures (i.e., mediport insertion), fine needle aspirates, or core biopsies within 7 days prior to the first date of bevacizumab/placebo therapy
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martee Hensley, Principal Investigator — NRG Oncology
Locations (201):
- United States (201):
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Rocky Mountain Gynecologic Oncology PC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mercy Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Georgia Regents University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cadence Cancer Center in Warrenville, Warrenville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Saint Francis Health-Indianapolis, Indianapolis, Indiana
  - Gynecologic Oncology of Indiana, Indianapolis, Indiana
  - Saint Vincent Oncology Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium CCOP, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Michiana Hematology Oncology PC-Niles, Niles, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota NCI Community Oncology Research Program, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin

REFERENCES:
- [Derived] Kantidakis G, Litiere S, Neven A, Vinches M, Judson I, Schoffski P, Wardelmann E, Stacchiotti S, D'Ambrosio L, Marreaud S, van der Graaf WTA, Kasper B, Fiocco M, Gelderblom H. Efficacy thresholds for clinical trials with advanced or metastatic leiomyosarcoma patients: A European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group meta-analysis based on a literature review for soft-tissue sarcomas. Eur J Cancer. 2021 Sep;154:253-268. doi: 10.1016/j.ejca.2021.06.025. Epub 2021 Jul 20. PMID 34298376
- [Derived] Hensley ML, Miller A, O'Malley DM, Mannel RS, Behbakht K, Bakkum-Gamez JN, Michael H. Randomized phase III trial of gemcitabine plus docetaxel plus bevacizumab or placebo as first-line treatment for metastatic uterine leiomyosarcoma: an NRG Oncology/Gynecologic Oncology Group study. J Clin Oncol. 2015 Apr 1;33(10):1180-5. doi: 10.1200/JCO.2014.58.3781. Epub 2015 Feb 23. PMID 25713428
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I Gem+Doce+Placebo | Arm II Gem+Doce+Bev
Started | 54 | 53
Completed | 54 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I Gem+Doce+Placebo | Arm II Gem+Doce+Bev | Total
Number analyzed (Participants) | 54 | 53 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (8.1) | 54.0 (8.7) | 55.7 (8.6)
Age, Customized [Count of Participants; unit: Participants]
  Age Groups: 20-29 years | 0 | 1 | 1
  Age Groups: 30-39 years | 0 | 3 | 3
  Age Groups: 40-49 years | 11 | 12 | 23
  Age Groups: 50-59 years | 24 | 25 | 49
  Age Groups: 60-69 years | 19 | 12 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 53 | 107
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 48 | 43 | 91
  Unknown or Not Reported | 2 | 7 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 12 | 18
  White | 46 | 36 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Prior whole pelvic radiation [Count of Participants; unit: Participants]
  Yes | 11 | 11 | 22
  No | 43 | 42 | 85
Performance Status [Count of Participants; unit: Participants]
  0: Asymptomatic | 38 | 41 | 79
  1: Symptomatic, fully ambulatory | 15 | 11 | 26
  2: Symptomatic, in bed < 50% of time | 1 | 1 | 2
FIGO Stage [Count of Participants; unit: Participants] — FIGO Stage describes disease burden at time of surgery. Stage 1 indicates the cancer has not spread beyond the uterus. Stage 4 indicates cancer metastasis in distant organs.
  Participants
    1 | 20 | 11 | 31
    2 | 4 | 0 | 4
    3 | 3 | 5 | 8
    4 | 22 | 30 | 52
    unknown | 5 | 7 | 12
Cell Type [Count of Participants; unit: Participants]
  Leiomyosarcoma | 52 | 52 | 104
  Sarcoma, Unsp. | 1 | 0 | 1
  Carcinsarcoma | 0 | 1 | 1
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression free survival (PFS) was defined as the number of months between study enrollment and documentation of disease progression (RECIST 1.1) or death from any cause. Patients still alive and disease free at the last followup were censored on the date of last CT Scan.
  Assessed with a log-rank test stratified by whether the patient had whole pelvic radiotherapy prior to starting the study treatment. The product-limit method will be used to estimate the cumulative distribution of PFS for the patients assigned to each treatment group.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Population: All randomized
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I Gem+Doce+Placebo | Arm II Gem+Doce+Bev
Number analyzed (Participants) | 54 | 53
months | 6.2 [2.9 to 9.9] | 4.2 [3.1 to 8.4]

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the number of months between study enrollment and death from any cause. Patients still alive at the last followup were censored on the date of last CT Scan.
  The product-limit method will be used to estimate the cumulative distribution of overall survival times for the patients assigned to each treatment group.
Time Frame: Up to 5 years
Population: All randomized
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I Gem+Doce+Placebo | Arm II Gem+Doce+Bev
Number analyzed (Participants) | 54 | 53
months | 26.9 [15.9 to 32.1] | 23.3 [16.6 to 27.3]

3. Secondary Outcome: Frequency and Severity of Adverse Effects as Assessed by the CTCAE Version 4.0
Description: Count of participants with Adverse events (AEs) that are CTCAE Grade 3 or worse.
  Please refer to the adverse event reporting for more detail.
Time Frame: Up to 5 years
Population: All randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Gem+Doce+Placebo | Arm II Gem+Doce+Bev
Number analyzed (Participants) | 54 | 53
Participants | 36 | 46

4. Secondary Outcome: Objective Response Rate as Measured by RECIST 1.1 Criteria
Description: "Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Population: All randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I Gem+Doce+Placebo | Arm II Gem+Doce+Bev
Number analyzed (Participants) | 54 | 53
percentage of participants | 31.5 [21.2 to 43.4] | 35.8 [24.9 to 48.0]

ADVERSE EVENTS:
Groups:
- Arm I: Patients receive a placebo IV over 30-90 minutes on day 1, gemcitabine hydrochloride IV over 90 minutes on days 1 and 8, and docetaxel IV over 60 minutes on day 8. Patients also receive filgrastim subcutaneously (SC) on days 9-15 or pegfilgrastim SC on day 9 or 10.
  Docetaxel: Given IV
  Filgrastim: Given SC
  Gemcitabine Hydrochloride: Given IV
  Pegfilgrastim: Given SC
  Placebo: Given IV
- Arm II: Patients receive bevacizumab IV over 30-90 minutes on day 1, gemcitabine hydrochloride IV over 90 minutes on days 1 and 8, and docetaxel IV over 60 minutes on day 8. Patients also receive filgrastim SC on days 9-15 or pegfilgrastim SC on day 9 or 10.
  Bevacizumab: Given IV
  Docetaxel: Given IV
  Filgrastim: Given SC
  Gemcitabine Hydrochloride: Given IV
  Pegfilgrastim: Given SC
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 17/54 | 21/53
Other Adverse Events (participants affected / at risk) | 51/54 | 51/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=54) | Arm II (N=53)
Pericardial Effusion (Cardiac disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 2 | 0
Anaphylaxis (Immune system disorders) | 0 | 1
Allergic Reaction (Immune system disorders) | 1 | 0
Infections And Infestations - Other (Infections and infestations) | 0 | 2
Soft Tissue Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 3 | 2
Catheter Related Infection (Infections and infestations) | 1 | 2
Abdominal Infection (Infections and infestations) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 3
Lymphocyte Count Decreased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thromboembolic Event (Vascular disorders) | 2 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=54) | Arm II (N=53)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 | 2
Anemia (Blood and lymphatic system disorders) | 47 | 48
Palpitations (Cardiac disorders) | 2 | 3
Pericardial Effusion (Cardiac disorders) | 1 | 1
Sinus Tachycardia (Cardiac disorders) | 3 | 5
Chest Pain - Cardiac (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Hearing Impaired (Ear and labyrinth disorders) | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 1 | 4
Eye Disorders - Other (Eye disorders) | 1 | 2
Watering Eyes (Eye disorders) | 1 | 9
Eye Pain (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 1
Blurred Vision (Eye disorders) | 6 | 4
Dry Eye (Eye disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 3
Dry Mouth (Gastrointestinal disorders) | 1 | 5
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 24 | 26
Diarrhea (Gastrointestinal disorders) | 19 | 22
Vomiting (Gastrointestinal disorders) | 14 | 16
Bloating (Gastrointestinal disorders) | 1 | 3
Stomach Pain (Gastrointestinal disorders) | 1 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Anal Hemorrhage (Gastrointestinal disorders) | 1 | 2
Rectal Fistula (Gastrointestinal disorders) | 0 | 1
Rectal Mucositis (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 16 | 15
Rectal Hemorrhage (Gastrointestinal disorders) | 5 | 2
Oral Dysesthesia (Gastrointestinal disorders) | 2 | 1
Mucositis Oral (Gastrointestinal disorders) | 14 | 15
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1 | 3
Oral Hemorrhage (Gastrointestinal disorders) | 0 | 4
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 1
Gingival Pain (Gastrointestinal disorders) | 1 | 1
Oral Pain (Gastrointestinal disorders) | 2 | 3
Abdominal Distension (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 35 | 29
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 6
Rectal Pain (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 3 | 3
Hemorrhoids (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Esophageal Pain (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
General Disorders And Administration Site Conditio (General disorders) | 2 | 0
Pain (General disorders) | 13 | 9
Localized Edema (General disorders) | 0 | 1
Injection Site Reaction (General disorders) | 2 | 2
Infusion Site Extravasation (General disorders) | 1 | 0
Flu Like Symptoms (General disorders) | 2 | 2
Edema Trunk (General disorders) | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 4 | 3
Edema Limbs (General disorders) | 23 | 12
Edema Face (General disorders) | 4 | 3
Fatigue (General disorders) | 45 | 42
Fever (General disorders) | 17 | 19
Chills (General disorders) | 3 | 3
Infusion Related Reaction (General disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Allergic Reaction (Immune system disorders) | 7 | 1
Cytokine Release Syndrome (Immune system disorders) | 1 | 0
Infections And Infestations - Other (Infections and infestations) | 2 | 1
Upper Respiratory Infection (Infections and infestations) | 2 | 1
Tooth Infection (Infections and infestations) | 1 | 3
Skin Infection (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 1
Papulopustular Rash (Infections and infestations) | 1 | 0
Nail Infection (Infections and infestations) | 1 | 3
Mucosal Infection (Infections and infestations) | 3 | 1
Pelvic Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 2 | 2
Eye Infection (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 2 | 1
Vaginal Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 8 | 7
Catheter Related Infection (Infections and infestations) | 0 | 2
Bronchial Infection (Infections and infestations) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Bladder Infection (Infections and infestations) | 0 | 1
Lip Infection (Infections and infestations) | 1 | 0
Anorectal Infection (Infections and infestations) | 0 | 1
Injury, Poisoning And Procedural Complications - O (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 1
Tracheostomy Site Bleeding (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 4
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Investigations - Other (Investigations) | 2 | 0
Weight Loss (Investigations) | 4 | 6
Weight Gain (Investigations) | 4 | 5
Platelet Count Decreased (Investigations) | 39 | 45
Lymphocyte Count Decreased (Investigations) | 2 | 5
Inr Increased (Investigations) | 2 | 0
Creatinine Increased (Investigations) | 2 | 3
Neutrophil Count Decreased (Investigations) | 26 | 25
Blood Bilirubin Increased (Investigations) | 2 | 1
White Blood Cell Decreased (Investigations) | 28 | 33
Aspartate Aminotransferase Increased (Investigations) | 9 | 10
Alkaline Phosphatase Increased (Investigations) | 16 | 17
Alanine Aminotransferase Increased (Investigations) | 14 | 10
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2 | 1
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 8 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 4
Hypokalemia (Metabolism and nutrition disorders) | 8 | 8
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 12 | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 | 9
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 7
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 21 | 19
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 13 | 12
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 20
Musculoskeletal Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 2 | 2
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 13 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 9
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 1 | 1
Tremor (Nervous system disorders) | 1 | 0
Spasticity (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 21 | 19
Peripheral Motor Neuropathy (Nervous system disorders) | 3 | 3
Paresthesia (Nervous system disorders) | 2 | 3
Memory Impairment (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 17 | 14
Dysgeusia (Nervous system disorders) | 6 | 8
Sinus Pain (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 9 | 7
Ataxia (Nervous system disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 11 | 10
Depression (Psychiatric disorders) | 5 | 7
Anxiety (Psychiatric disorders) | 10 | 9
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 2 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 4
Urinary Tract Pain (Renal and urinary disorders) | 2 | 1
Urinary Frequency (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 2 | 1
Hemoglobinuria (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 2 | 2
Cystitis Noninfective (Renal and urinary disorders) | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 1
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 0 | 1
Vaginal Pain (Reproductive system and breast disorders) | 0 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 2 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 3
Breast Pain (Reproductive system and breast disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pharyngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 25
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 20
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 5 | 4
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 5
Rash Acneiform (Skin and subcutaneous tissue disorders) | 5 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Periorbital Edema (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 2
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 8 | 5
Nail Ridging (Skin and subcutaneous tissue disorders) | 1 | 1
Nail Loss (Skin and subcutaneous tissue disorders) | 3 | 3
Nail Discoloration (Skin and subcutaneous tissue disorders) | 2 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 7
Body Odor (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 36 | 34
Vascular Disorders - Other (Vascular disorders) | 0 | 1
Thromboembolic Event (Vascular disorders) | 6 | 4
Superficial Thrombophlebitis (Vascular disorders) | 0 | 1
Lymphedema (Vascular disorders) | 0 | 4
Hypotension (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 10 | 12
Hot Flashes (Vascular disorders) | 2 | 7
Hematoma (Vascular disorders) | 1 | 1
Flushing (Vascular disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
The study was targeted to accrue 130 patients, but closed early for futility. Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less